CLINICAL TRIAL: NCT06058195
Title: Comparison of the Efficacy of Bilateral Transverse Abdominis Plane Block (TAPB) and Bilateral Quadratus Lumborum Block (QLB) With Intravenous Analgesic (IVA) Group for Preemptive Analgesia in Laparoscopic Cholecystectomy Surgery
Brief Title: Comparison of Quadratus Lumborum and Transverse Abdominis Plane Blocks With Intravenous Analgesic in Gallbladder Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 03.03.2023/372
Record Dates: First submitted 2023-09-14; First posted 2023-09-28 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group QLB (quadratus lumborum plane block): Group QLB (quadratus lumborum plane block): 20 ml of 0.25% bupivacaine will be used each time for plane block on both sides. Patients will be sedated with 1 mg midazolam and 50 mcg fentanyl intravenously in the preoperative preparation room in the operating room and 20 ml of 0.25% bupivacaine was administered bilaterally on each side under ultrasound guidance. After the block application, the patient was taken to the operating room and standard general anaesthesia was applied.
  - Plane block applications will be applied only once in the preoperative period
  Interventions: Procedure: Quadratus lumborum plane block
- Group TAPB (transverse abdominis plane block): Group TAPB (transverse abdominis plane block): 20 ml of 0.25% bupivacaine will be used each time for plane block on both sides. Patients will be sedated with 1 mg midazolam and 50 mcg fentanyl intravenously in the preoperative preparation room in the operating room and 20 ml of 0.25% bupivacaine was administered bilaterally on each side under ultrasound guidance. After the block application, the patient was taken to the operating room and standard general anaesthesia was applied.
  Interventions: Procedure: Transverse abdominis plane block
- Group IVA (Intravenous analgesia): Group IVA (Intravenous analgesia): These patients will be administered 1000 mg paracetamol intravenously in the preoperative waiting room in the operating room approximately 20-30 minutes before induction of anaesthesia. No block procedure will be performed. Patients will not be given any analgesic medication before awakening from anaesthesia.
  Interventions: Procedure: Intravenous analgesia

INTERVENTIONS:
Procedure: Quadratus lumborum plane block — QLB (quadratus lumborum plane block): 20 ml of 0.25% bupivacaine will be used each time for plane block on both sides. Patients will be sedated with 1 mg midazolam and 50 mcg fentanyl intravenously in the preoperative preparation room in the operating room and 20 ml of 0.25% bupivacaine was administered bilaterally on each side under ultrasound guidance. After the block application, the patient was taken to the operating room and standard general anaesthesia was applied.
  Groups: Group QLB (quadratus lumborum plane block)
Procedure: Transverse abdominis plane block — TAPB (transverse abdominis plane block): 20 ml of 0.25% bupivacaine will be used each time for plane block on both sides. Patients will be sedated with 1 mg midazolam and 50 mcg fentanyl intravenously in the preoperative preparation room in the operating room and 20 ml of 0.25% bupivacaine was administered bilaterally on each side under ultrasound guidance. After the block application, the patient was taken to the operating room and standard general anaesthesia was applied.
  Groups: Group TAPB (transverse abdominis plane block)
Procedure: Intravenous analgesia — IVA (Intravenous analgesia): These patients will be administered 1000 mg paracetamol intravenously in the preoperative waiting room in the operating room approximately 20-30 minutes before induction of anaesthesia. No block procedure will be performed. Patients will not be given any analgesic medication before awakening from anaesthesia.
  Groups: Group IVA (Intravenous analgesia)

SUMMARY:
Patients who will undergo laparoscopic gallbladder surgery are expected to experience less postoperative pain and have less need for morphine-derived painkillers.

For this reason, a total of 128 patients were planned to be included in the study, including a group of patients who were eligible for gallbladder surgery with transverse abdominis plane block (TAPB), a group of patients with quadratus lumborum plane block (QLB) and a group of patients with intravenous painkillers (IVA).

DETAILED DESCRIPTION:
1. Group QLB (Quadratus lumborum plane block): 20 ml of 0.25% bupivacaine will be used each time for plane block on both sides. Patients will be sedated with 1 mg midazolam and 50 mcg fentanyl intravenously in the preoperative preparation room in the operating room and 20 ml of 0.25% bupivacaine was administered bilaterally on each side under ultrasound guidance. After the block application, the patient was taken to the operating room and standard general anaesthesia was applied. Patients will not be given any analgesic medication before awakening from anaesthesia.
2. Group TAPB (Transverse abdominis plane block): 20 ml of 0.25% bupivacaine will be used each time for plane block on both sides. Patients will be sedated with 1 mg midazolam and 50 mcg fentanyl intravenously in the preoperative preparation room in the operating room and 20 ml of 0.25% bupivacaine was administered bilaterally on each side under ultrasound guidance. After the block application, the patient was taken to the operating room and standard general anaesthesia was applied. Patients will not be given any analgesic medication before awakening from anaesthesia.

   For both Group QLB and Group TAPB block group;
   * Medical records will be audited to monitor adherence to the intervention.
   * each patient will be administered 0.25% bupivacaine for each side (a total of 40 ml of 0.25% bupivacaine will be used)
   * plane blocks will be applied under ultrasound guidance.
   * plane block applications will be performed by anaesthesiologists with at least 5 years of experience
   * Postoperative evaluations of patients will be performed face to face.
   * Plane block applications will be applied only once in the preoperative period.
   * In the postoperative period, 1000 mg paracetamol will be given intravenously if the pain intensity of the patients is below Visual Analogue Scale (VAS) 4. However, if the severity of pain is VAS 4 and above, 100 mg tramadol will be given intravenously.
   * This study will be followed up in the general surgery unit.
   * Patients will be monitored for pain and side effects at 30th minute, 2nd hour, 4th hour, 12th hour and 24th hour in the postoperative period.
   * Both plane blocks are applied for analgesia in the postoperative period and aim to reduce opioid consumption in the postoperative period.
3. Group IVA (Intravenous analgesia): These patients will be administered 1000 mg paracetamol intravenously in the preoperative waiting room in the operating room approximately 20-30 minutes before induction of anaesthesia. No block procedure will be performed. Patients will not be given any analgesic medication before awakening from anaesthesia.

   * Postoperative evaluations of patients will be performed face to face.
   * Plane block applications will be applied only once in the preoperative period.
   * In the postoperative period, 1000 mg paracetamol will be given intravenously if the pain intensity of the patients is below Visual Analogue Scale (VAS) 4. However, if the severity of pain is VAS 4 and above, 100 mg tramadol will be given intravenously.
   * This study will be followed up in the general surgery unit.
   * Patients will be monitored for pain and side effects at 30th minute, 2nd hour, 4th hour, 12th hour and 24th hour in the postoperative period.

Statistical methods / analysis: Power analysis (G-Power version 3.1.9.4 (University Kiel, Germany) program was used to calculate the sample size. The two-tailed alpha error was taken as 0.05, power as 0.80 and effect size as 0.8, and based on a previous study the allocation ratio was accepted as N2/N1:1. The minimum number of patients to be included in the study was calculated as 52.

SPSS 16.0 for Windows (SPSS Inc., Chicago, USA) was used for other statistical analyses. Statistical data were expressed as mean and standard deviation, while categorical data were expressed as frequency and percentage. Comparison of categorical data in the groups was done with Chi-square, the results were given as %n. Shapiro-Wilk tests were used to determine if the numerical data fit the normal distribution. While the data fitting the normal distribution were evaluated with the Student's t-test. Mann- Whitney U tests were used to compare the data differ from the normal distribution. p <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years,
* who will undergo laparoscopic cholecystectomy and who meet the American Society of Anesthesiologists (ASA) I-III physical status

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status above 3
* Age < 18 or >70 years
* patient's reluctance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo laparoscopic cholecystectomy surgery.
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-16 (Estimated)

PRIMARY OUTCOMES:
VAS value of abdominal pain | 30 minutes, 2 hours, 4 hours, 12 hours, 24 hours after the patient is extubated
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
postoperative total tramadol consumption | during the first 24 hours after surgery.
  Amount of tramadol used postoperatively (milligrams). If the VAS value of the patients is 4 and above, 100 mg tramadol is administered intravenously.

SECONDARY OUTCOMES:
Sedation- agitation level | during extubation
  The Richmond Agitation Sedation Scale (RASS): identifies seven levels of sedation and agitation, which range from dangerous agitation to deep sedation, with a thorough description of patient behavior.
  The Richmond Agitation Sedation Scale (RASS) is a 10-point scale ranging from -5 to +4.Levels -1 to -5 denote 5 levels of sedation, starting with "awakens to voice" and ending with "unarousable." Levels +1 to +4 describe increasing levels of agitation. The lowest level of agitation starts with apprehension and anxiety, and peaks at combative and violent. RASS level 0 is "alert and calm.
amount of fentanyl consumed during the operation | during surgery
  micrograms of fentanyl consumed during surgery
nausea-vomiting | 30 minutes, 2 hours, 4 hours, 12 hours, 24 hours after the patient is extubated
  questioning about the presence/absence of nausea and/or vomiting in the postoperative period
postoperative shoulder pain | 30 minutes, 2 hours, 4 hours, 12 hours, 24 hours after the patient is extubated
  shoulder pain patients will be asked to verbally assess whether there is pain or not
surgical duration | at the end of surgery
  Time in hours from the start of the surgical incision until the last surgical suture is placed
anaesthesia duration | at the end of anaesthesia
  time in hours from induction of anaesthesia to extubation
length of hospital stay | It is assessed for up to 12 months from the date of surgery to the date of the first documented progression or the date of death from any cause, whichever comes first
  days of hospitalisation after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Acil, Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Verma K, Malawat A, Jethava D, Jethava DD. Comparison of transversus abdominis plane block and quadratus lumborum block for post-caesarean section analgesia: A randomised clinical trial. Indian J Anaesth. 2019 Oct;63(10):820-826. doi: 10.4103/ija.IJA_61_19. Epub 2019 Oct 10. PMID 31649394